CLINICAL TRIAL: NCT03327753
Title: Which Exercise for Low Back Pain? Predicting Response to Exercise Treatments for Patients With Low Back Pain: a Validation Pilot Study
Brief Title: Which Exercise for Low Back Pain: A Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Alberta (Other); Macquarie University, Australia (Other)
Responsible Party: Principal Investigator, Luciana Macedo, Assistant Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WhichEx2017
Record Dates: First submitted 2017-10-23; First posted 2017-10-31 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Chronic Low Back Pain; Non Specific Low Back Pain
Keywords: exercise; mobility; physiotherapy; validation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into one of two groups, both of which are exercises considered part of standard care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given that this is an exercise study blinding of participants and those delivering the exercise program will not be possible. Outcome measures will be collected by an investigator not aware of treatment allocation, but most outcome measures will be self-reported and thus, true assessor blinding will no be possible. All statistical analysis will be conducted by a blinded investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor control exercises (Experimental): A primary goal of the motor control exercise program is to regain control and coordination of the spine and pelvis using principles of motor learning such as segmentation and simplification. The whole intervention is based on assessment of the individual patient's motor control impairments and the patient's individual treatment goals (set collaboratively with the therapist).
  Interventions: Behavioral: Motor control exercises
- Graded activity (Experimental): A primary goal of the graded activity program is to increase activity tolerance by performing individualized and submaximal exercises in addition to ignoring illness behaviors and reinforcing well behaviors. The intervention uses cognitive behavioral approaches to deal with fear of movement and self efficacy.
  Interventions: Behavioral: Graded activity

INTERVENTIONS:
Behavioral: Motor control exercises — The first stage of the treatment involves assessment of symptoms and implementation of a retraining program designed to improve activity of muscles assessed to have poor control and reducing activity of any muscle identified to be overactive. Participants are taught how to contract these muscles independently from the superficial trunk muscles and progress until the patient are able to maintain isolated contractions of the target muscles. During this stage exercises for breathing control, posture of spine and lower limb and movement are performed. The second stage of the treatment involved the progression of the exercises towards more functional activities. Throughout this process the recruitment of the trunk muscles, posture, movement pattern and breathing are assessed and corrected.
  Arms: Motor control exercises
Behavioral: Graded activity — The program is based on activities that each patient identify as problematic and that they cannot perform or have difficulty performing because of their back pain. The activities in the program are progressed in a time-contingent manner from the baseline assessed ability to a target goal set jointly by patient and therapist. Patients receive daily quotas and are instructed to only perform the agreed amount, even when they feel they are capable of doing more. Cognitive-behavioural principles are used to help patients overcome the natural anxiety associated with pain and activities. Physiotherapists use positive reinforcement, explain pain mechanisms and addressed negative behaviours and pain-related anxiety. A plan for managing relapses is developed between therapists and patients.
  Arms: Graded activity

SUMMARY:
Dr. Macedo and others involved in the proposed research recently conducted a study that investigated whether simple clinical characteristics could identify patients who benefit more from either motor control exercises or graded activity. Results were statistically significant and clinically relevant demonstrating that a simple questionnaire could help aid the selection of the most appropriate exercise therapy for each individual patient. Therefore, we aim to conduct a randomized controlled trial following a similar approach to the original study to validate in a different sample the results of the effect modification analysis.

DETAILED DESCRIPTION:
Dr. Macedo and others involved in the proposed research recently conducted a study that investigated whether simple clinical characteristics could identify patients who benefit more from either motor control exercises or graded activity. Motor control exercises (sometimes called lumbar stabilization exercises) and graded activity using the principles of cognitive behavioral therapy are two popular forms of exercise therapy with evidence of effectiveness from high quality systematic reviews, but no evidence for superiority of one approach over the other when tested in heterogenous populations. The results of a previously published study demonstrated that a simple 15-item questionnaire (Lumbar Spine Instability (LSI) Questionnaire) could identify patients who responded best to either motor control exercise or graded activity (interaction 2.72 95% CI 1.39 to 4.06, p=0.001). The results demonstrated that for people who are LSI negative, graded activity provided a much better outcome than motor control exercise one year post-intervention (a statistically and clinically significant improvement of 1.96 points on a 0-10 numeric function scale; p< 0.001). In people who were LSI positive, motor control exercise provided slightly better outcomes, compared to those prescribed motor control exercises. It is important to note that this study was measuring differences between treatments groups, and thus change in the scores of function presented represent differences between groups.

However, although this clinical decision rule has the potential to transform exercise treatment for LBP, especially given the relatively large interaction effects found, validation in an independent sample is essential before recommending use in clinical practice.There are three recognized steps in developing clinical decisions rules: derivation, validation and impact evaluation. Dr. Macedo's previous study falls within the first step of this process and the proposed study aims to address the second step; validation.

Therefore, the objective of this study is to conduct a randomized controlled trial following a similar approach to the original study to validate in a different sample the results of the effect modification analysis to identify baseline characteristics that predict/modify response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible for inclusion if they meet all of the following inclusion criteria: chronic non-specific LBP (>3 months) with or without leg pain, currently seeking care for LBP, between 18 to 80 years of age, English speaking (to allow response to the questionnaires and communication with the treating physiotherapist), Clinical assessment indicating that the participant is suitable for active exercises (by a family physician or using the Physical Activity Readiness Questionnaire), Moderate or greater pain or disability measured using question 7 or question 8 of the SF-36 Health Survey, moderate or High Risk Classification on the STarT Back Tool indicating appropriateness of physiotherapy and thus an exercise program.

Exclusion Criteria:

* Exclusion criteria will be known or suspected serious pathology, comorbidity that would prevent participation in exercise programs and scheduled for surgery during trial period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Patient Specific Functional Scale | 12 months
  This scale evaluates patient's self function on a scale from 0-10.

SECONDARY OUTCOMES:
Patient Specific Functional Scale | 2 and 6 month
  This scale evaluates patient's self reported function on a scale from 0-10
Roland Morris Disability Questionnaire | 2, 6 and 12 months
  The RMDQ questionnaires evaluates pain related disability on a scale from 0-24.
Numeric Rating Scale- pain | 2, 6 and 12 months
  A numeric rating scale from 0-10 will be used to assess average level of pain over the last week
SF-36 | 2, 6 and 12 months
  The SF-36 will be used to assess self reported quality of life

OTHER OUTCOMES:
Effect Modifier - OREBRO | baseline
  OREBRO LBP screening questionnaire is a 24 item scale to measure psychosocial risk factors for poor outcomes (scale from 11 to 192)
Effect modifier _ Lumbar instability | baseline
  Lumbar Spine Instability Questionnaire is a self reported scale to evaluate clinical instability on a scale from 0-15.
Effect modifier _ Kinesiophobia | baseline
  Pain Anxiety Symptom Scale (PASS - 20) is a scale used in chronic pain to evaluate kinesiophobia, anxiety and depression symptoms associated with pain experience. Scores are divided into cognitive (0 to 5), escape/avoidance (0 to 5), fear (0 to 5) and psychological anxiety (0 to 5). Total score from 0-100
Effect modifier_ Coping | baseline
  Coping Strategies Questionnaire is a 6 item measure of coping in patients with chronic pain (00-36)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Macedo, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No